CLINICAL TRIAL: NCT06690073
Title: The Effect of Motor Relearning Program on Functional Mobility in Stroke Rehabilitation
Acronym: MRP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Collaborators: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Karthick Balasubramanian, Lecturer, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Apr.13/COM-2022/32-3
Record Dates: First submitted 2024-11-10; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Chronic Stroke Patients; Chronic Stroke Survivors; Hemiplegia
Keywords: Stroke; Hemiplegia; Functional mobility; motor relearning program
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Conventional Physical Therapy (CPT) was administered to the control group three times per week for six weeks (45 minutes per session). CPT treatments such as mat activities, assisted movements, weight-bearing strategies, and gymnasium training were given to the control group.
  Interventions: Other: Conventional Physical Therapy
- Experimental (Experimental): the experimental group received the previously mentioned CPT treatment as well as MRP for sitting to standing for six weeks, for a total duration of 45 minutes per session (30 minutes of CPT treatment followed by 15 minutes MRP), three sessions per week.
  MRP of sitting and standing activities: The physical therapist was standing in front of the participant, who was sitting in an armrest-equipped chair. Participants were initially taught to keep their feet back, followed by forward trunk positioning. The physical therapist then aided the activity by holding the involved side of the hand and shoulder, where the subject had informed to execute anterior trunk bending more quickly, if the participant did not do it well or performed it in an abnormal manner. Finally, participants were instructed to press down through the affected foot, stand up as quickly as possible, and bring their hips anterior. The physical therapist suggested pressing down through the participant's knee along the shaft
  Interventions: Other: Motor Relearning Program

INTERVENTIONS:
Other: Motor Relearning Program — Total duration of the intervention is 45 minutes per session (30 minutes of CPT treatment followed by 15 minutes MRP), three sessions per week.
  MRP of sitting and standing activities: The physical therapist will instruct the participant, who will be seated in an armrest-equipped chair, to keep their feet back and position their trunk forward.. The participant will then be guided to press down through the affected foot, stand up quickly, and move their hips forward. The therapist will suggest pressing down through the participant's knee along the leg while moving it forward through the affected foot.
  MRP of standing to sitting: The participant will stand while the physiotherapist assists with anterior shoulder movement and knee bending at the start of the transition. The therapist will then help maintain weight on the affected leg while sitting. The participant will progress by standing and sitting at different seat heights, stopping at various points in the ROM, and changing speed.
  Other Names: Conventional Physical Therapy
  Arms: Experimental
Other: Conventional Physical Therapy — Conventional Physical Therapy (CPT) will be administered to the control group three times per week for six weeks (45 minutes per session). CPT treatments such as mat activities, assisted movements, weight-bearing strategies, and gymnasium training will be given to the control group.
  Arms: Control

SUMMARY:
1. To find out the effectiveness of conventional physiotherapy on improving functional mobility of lower extremity among chronic hemiplegic subjects.
2. To find out the effcctiveness of motor relearning program along with conventional physical therapy treatment on improving functional mobility of lower extremity among chronic hemiplegic subjects.
3. To find out the effectiveness of motor relearning program along with conventional physical therapy treatment over conventional physical therapy on improving functional mobility of lower extremity among chronic hemiplegic subjects.

DETAILED DESCRIPTION:
After a careful monitor of inclusion and exclusion criteria and obtaining the institutional review board approval, the study was conducted by convenience sampling to select the suitable subjects, explaining the procedure to them, and got the written & oral informed consent. The study included two groups, each with 16 participants, which were allocated randomly to the control and experimental groups by lottery method. CPT was administered to the control group three times per week for six weeks (45 minutes per session). CPT treatments such as mat activities, assisted movements, weight-bearing strategies, and gymnasium training were given to the control group. At the same time, the experimental group received the previously mentioned CPT treatment as well as MRP for sitting to standing for six weeks, for a total duration of 45 minutes per session (30 minutes of CPT treatment followed by 15 minutes MRP), three sessions per week.

MRP of sitting and standing activities: The physical therapist was standing in front of the participant, who was sitting in an armrest-equipped chair. Participants were initially taught to keep their feet back, followed by forward trunk positioning. The physical therapist then aided the activity by holding the involved side of the hand and shoulder, where the subject had informed to execute anterior trunk bending more quickly, if the participant did not do it well or performed it in an abnormal manner. Finally, participants were instructed to press down through the affected foot, stand up as quickly as possible, and bring their hips anterior. The physical therapist suggested pressing down through the participant's knee along the shaft of the leg while moving it anteriorly through the affected foot.

MRP of standing to sitting: The participant was on his feet. The physiotherapist assisted the participant with anterior shoulder movement and knee bending at the start of the stand-to-sit movement. The physiotherapist then assisted the participant in keeping his weight on the affected leg while sitting. The subject progressed by standing and sitting with different seat heights, stopping in different parts of the range of motion, and varying speed. These variations in time and space were directed by the physical therapist. The number of reps and intensity of the exercise were classified according to the subject's capacity level and gradually increased as they improved. Subjects were given verbal feedback on weight distribution, performance speed, and encouragement.

ELIGIBILITY:
Inclusion criteria: The following subjects were included:

* Right or left-sided chronic hemiplegic subjects.
* More than six months after the onset of stroke.
* Age group between 45-65 years of both genders.
* Scored minimally 24/30 on the Mini-Mental State Exam (MMSE).
* Motor assessment scale of sitting to standing section.
* Having normal visual perception.
* Able to follow verbal commands.

Exclusion criteria: The following subjects were excluded:

* Less than six months after the onset of stroke.
* Unable to follow visual and oral commands.
* The age group is below 45 years and more than 65 years.
* Unilateral neglect.
* Cognitive impairments (MMSE scores less than 24/30), or language deficits.
* Any other neurological disorders and recent surgeries.
* Previous exposure to MRP.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Barthel Index (BI) | week 0 and week 6
  The Barthel index, frequently used for stroke, gauges the level of help needed by an individual for ten mobility and daily living tasks. The total of all weighted individual item scores is converted into a single overall score, which ranges from 0 to 100. Consequently, "0" represents total independence from all ten activities. It takes 5 to 10 minutes to complete, has strong validity and reliability, and has minimal sensitivity for high-level functioning (Bhalerao et al., 2011).
Motor Assessment Scale (MAS) | week 0 and week 6
  MAS is used to evaluate motor skills. MAS records eight functional activities: rolling in bed, sitting, sit to stand, walking, balancing in seated position, upper arm, hand, and wrist activities. The general tone of the body is noted in the ninth item. The scale for each item is 0 to 6. Hence, a score of 0 to 54 (normal function). According to WHO guidelines, MAS is supposed to be tested on the severity of disabilities. The MAS was highly dependable, with an average inter-rater reliability of .95 and an average test-retest reliability of 0.98 (Bhalerao et al., 2011).

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud Medical City, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alfaleh KA, Shaik AR, Balasubramanian K, Alshehri MM, Sanjeevi RR, Esht V, Alsalem WO, Shahhar AM, Alothman SA. Effectiveness of motor relearning program in sit-to-stand transfer and activities of daily living among chronic stroke patients - a prospective, multicenter, randomized controlled trial. J Comp Eff Res. 2026 Jan;15(1):e250133. doi: 10.57264/cer-2025-0133. Epub 2025 Dec 9. PMID 41363941